CLINICAL TRIAL: NCT06716385
Title: A Prospective, Randomized, Double-blind, Parallel, Active-controlled Clinical Trial to Evaluate the Vision Correction Safety and Efficacy of MSiHy Silicone Hydrogel Soft Contact Lens
Brief Title: A Clinical Trial to Evaluate the Vision Correction Safety and Efficacy of MSiHy Silicone Hydrogel Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visco Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0474TC01
Record Dates: First submitted 2024-08-28; First posted 2024-12-04 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Refractive Errors
Keywords: Contact lens
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- MSiHy Silicone Hydrogel Soft Contact Lens (Experimental): New Monthly disposable contact lenses
  Interventions: Device: MSiHy Silicone Hydrogel Soft Contact Lens
- Monthly Silicone Hydrogel Contact Lenses (oA) (Active Comparator): Monthly disposable contact lens products already on the market
  Interventions: Device: Monthly Silicone Hydrogel Contact Lenses (oA)

INTERVENTIONS:
Device: MSiHy Silicone Hydrogel Soft Contact Lens — The daily wear, monthly disposable soft contact lens for the correction of myopia and hyperopia in person with non-diseased eyes.
  Arms: MSiHy Silicone Hydrogel Soft Contact Lens
Device: Monthly Silicone Hydrogel Contact Lenses (oA) — The daily wear, monthly disposable soft contact lens for the correction of myopia and hyperopia in person with non-diseased eyes.
  Arms: Monthly Silicone Hydrogel Contact Lenses (oA)

SUMMARY:
This is a prospective, randomized, double-blind, parallel, active-controlled, multi-center clinical study. The purpose is to evaluate the safety and effectiveness wearing "MSiHy Silicone Hydrogel Soft Contact Lens".

Subjects will be randomized in 1:1 ratio to wear either the investigational device "MSiHy Silicone Hydrogel Soft Contact Lens" or the control device Monthly Silicone Hydrogel Contact Lenses(oA)".

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age inclusive
2. Beside myopia and astigmatism, subjects with normal eyes and are not using any ocular medications (excluding ocular lubricants and artificial tears)
3. Best spectacle corrected visual acuity greater than or equal to 1.0 for both eyes
4. With +8.00D ~ -12.00 D spherical component myopia, and ≤1.00 astigmatism (based on manifest refraction measurements)
5. Have worn soft contact lens for at least 2 month prior to the study
6. Willing to comply with the required wearing time
7. Agree to comply with all study procedures, sign and date the informed consent form before starting the clinical study

Exclusion Criteria:

1. Anterior segment infection, inflammation or abnormality
2. Any active ocular disease that would affect contact lens wear or vision (such as acute and subacute inflammation of the anterior chamber of the eye, eye infection, uveitis, serious palpebral abnormality, corneal hypoesthesia, corneal epithelium abrasion, dry eye and tear duct defection, ocular allergies, highly suspected glaucoma) upon evaluation by the investigators or slit lamp findings
3. Currently using systemic or ocular medications that would contraindicate contact lens wear (such as glaucoma eye drops, steroid anti-inflammatory drops, eye ointments, eye gels and other eye medicines)
4. History of herpetic keratitis
5. History of refractive surgery, keratoconus or irregular cornea
6. Slit lamp findings that are not suitable for inclusion (Details of the grading standards for each eye condition are specified in CIP section 5.7.5)
7. A pathologically dry eye (Schirmer test 1 <5 mm)
8. Have participated in any contact lens or contact lens care product clinical trials within the previous 1 month (excluding questionnaire types and specimen collection)
9. Currently pregnant, lactating, or planning to be pregnant during the trial
10. Have experienced discomfort when wearing silicone hydrogel contact lens, or a known allergy to hyaluronic acid and sodium alginate
11. Allergy to any contact lens care product ingredient
12. Corrected visual acuity in either eye does not reach 1.0 when wearing the trial lens
13. Subjects who are judged by the investigators as unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Visual Correction | 3 months
  The effectiveness of vision correction is defined by the proportion of subjects whose contact lens corrected visual acuity in both eyes is 1.0 or greater.

SECONDARY OUTCOMES:
Visual Correction | 1 week, 2 week, 1 month and 2 months
  The effectiveness of vision correction is defined by the proportion of subjects whose contact lens corrected visual acuity in both eyes is 1.0 or greater.
Change in refraction | 1 week, 2 week, 1 month, 2 months and 3 months
  the sphere and cylinder power of subjective refraction

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - MayKay Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No